CLINICAL TRIAL: NCT05403294
Title: Impact of New Anthropometric Indices on Outcomes After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, MERVE SAHINGOZ, Principal Investigator, TC Erciyes University
Other Study IDs: 2022/02
Record Dates: First submitted 2022-05-02; First posted 2022-06-03 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease; Cardiometabolic Risk Factors; Cardiac Anesthesia; Cardiac Surgery; Anthropometry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is associated with a number of risk factors for cardiovascular disease. Body mass index (BMI) is the most commonly recommended and used anthropometric measure to classify general obesity in clinical and epidemiological studies. It is widely accepted that obesity increases the risk of heart disease and is thought to be a risk factor for adverse outcomes after cardiac surgery. However, recent studies show paradoxical results, wherein obese patients can experience fewer adverse events and lower mortality than patients with normal-low body mass index(BMI) . The discriminative capacity of BMI has been criticized because it cannot distinguish muscle mass from fat mass, or reflect fat distribution . Alternatively, abdominal obesity indices, such as waist circumference (WC) and waist-to-height ratio (WHtR), have been suggested to be better predictor of cardiometabolic abnormalities because they modulate the limitation of BMI. However, they were insufficient in studies.For this reason, scientists turned to find a new anthropometric formula that could better detect obesity-related mortality and morbidity and they developed 2 new methods. Body Shape İndex (ABSI) is calculated using waist circumference, BMI and height parameters. Body Roundness İndex (BRI) is calculated using waist circumference and height parameters. These new indices may reflect visceral adiposity and strongly predict cardiovascular risk, postsurgical outcomes and resource utilisation.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery
* voluntary patients

Exclusion Criteria:

* emergency surgery
* off-pump or robotic surgery
* surgery requiring deep hypothermic circulatory arrest
* reluctant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who have undergone open heart surgery
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-07-27 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
mortality | within 30 days of the procedure
  Number of death at 30 days after surgery
postoperative stroke | within 30 days of the procedure
  Number of patients with postoperative stroke
cardiac arrest | within 30 days of the procedure
  number of patients with cardiac arrest
new atrial fibrillation/flutter | within 30 days of the procedure
  Number of Partients with new atrial fibrillation/flutter
permanent rhythm device insertion | within 30 days of the procedure
  Number of Patients requiring insertion of a permanent device

SECONDARY OUTCOMES:
prolonged ventilation | within 30 days of the procedure
  number of patients experiencing prolonged postoperative pulmonary ventilation (>24 hours)
sepsis /deep sternal infection | within 30 days of the procedure
  number of patients with sepsis, deep sternal wound infection or mediastinitis
pulmonary complications | within 30 days of the procedure
  number of patients with pneumonia or pleural effusion
renal failure / renal dialysis | within 30 days of the procedure
  number of patient with acute renal failure or worsening renal function result
total intensive care unit (ICU) hours | within 30 days of the procedure
  total intensive care unit (ICU) hours
intensive care unit (ICU) readmissions | within 30 days of the procedure
  number of patients with intensive care unit readmission